CLINICAL TRIAL: NCT07276555
Title: Efficacy and Safety of Functional Neurogenesis Stimulation Therapy in Children With Autism Spectrum Disorder: A Multicenter, Randomized Controlled Trial
Brief Title: Efficacy and Safety of Functional Neurogenesis Stimulation Therapy in Children With Autism Spectrum Disorder (ASD)
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Neurocytonix, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NCX-ASD-02
Record Dates: First submitted 2025-11-29; First posted 2025-12-11 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-12

CONDITIONS: Autism Spectrum Disorder
Keywords: Neurocytotron; Autism Spectrum Disorder; ASD; Functional Neurogenesis Stimulation Therapy
MeSH Terms: conditions — Autism Spectrum Disorder

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- Placebo Control Group (Placebo Comparator): Group not treated with Functional Neurogenesis Stimulation Therapy (NeuroCytotron)
  Interventions: Other: placebo control group
- Functional Neurogenesis Stimulation Therapy Treatment Group (Experimental): Group treated with Functional Neurogenesis Stimulation Therapy (NeuroCytotron)
  Interventions: Device: Functional Neurogenesis Stimulation Therapy

INTERVENTIONS:
Device: Functional Neurogenesis Stimulation Therapy — NeuroCytotron is a noninvasive investigational medical device that delivers Functional Neurogenesis Stimulation using low-energy, pulsed electromagnetic fields to specific brain regions. For this study, each participant receives one 60-minute treatment session per day for 28 consecutive days. Treatment parameters (field strength, frequency, and beam geometry) are individualized for each child based on their baseline brain MRI to define a three-dimensional target volume. During each session, the child sits or lies comfortably inside the device while the pre-programmed treatment plan is delivered; no surgery, implants, or systemic medications are used.
  Other Names: NeuroCytotron
  Arms: Functional Neurogenesis Stimulation Therapy Treatment Group
Other: placebo control group — This group will be placed on the device, but will not be treated (placebo group).
  Arms: Placebo Control Group

SUMMARY:
This study will test whether a noninvasive brain stimulation treatment called Functional Neurogenesis Stimulation (using the NeuroCytontron device) can safely improve core symptoms of Autism Spectrum Disorder (ASD) in children. The study will enroll boys and girls 3 to 12 years old who have ASD (DSM-5 level 1 - 2) and use at least some spoken language. Children may be randomly assigned (like a coin flip) to receive either active NeuroCytotron sessions or sham (placebo) sessions that look the same but deliver no active treatment. Neither the families nor the study staff doing the assessments will know which treatment a child is receiving. The primary question is whether children who receive active treatment exhibit greater improvement in social communication, interaction, and repetitive behaviors compared to children who receive a placebo, as measured by standard autism rating scales.

Each child's participation will last about 3 to 4 months, including screening, 28 days of daily, 1-hour treatment sessions, and follow-up visits up to 12 weeks after the last treatment. During the study, children will undergo physical exams, vital sign assessments, blood and urine tests, brain MRI scans, and electroencephalogram (EEG) recordings to examine brain structure and activity. Some children may need mild sedation or anesthesia for an MRI, which has its own risks. The device utilizes low-energy electromagnetic fields, similar to those used in MRIs. Possible risks include discomfort from lying still, anxiety around the device or MRI scanner, and side effects from sedation or from unexpected changes in behavior or seizures. There may or may not be direct benefit to each child, but information from this study may help researchers develop new, noninvasive treatment options for children with ASD in the future.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects with a confirmed diagnosis of ASD according to DSM-5
* criteria.
* Subjects ≥ 3 and ≤ 12 years.
* Subjects with ASD severity grade 1 to 2 according to DSM-5 criteria.
* Participants must have functional use of language (i.e., at least some verbal
* communication) to ensure that they engage with the assessments.
* Stable on current medications for at least 4 weeks prior to the study.
* To have the informed consent of the parents or legal representatives for the subject's
* participation in the study.
* Subjects must be physically able and willing to undergo the treatment sessions.
* Subjects must be medically and psychologically stable to participate in the study.

Exclusion Criteria:

* Presence of medical conditions that could contraindicate the use of NeuroCytotron,
* such as severe neurological disorders and difficult-to-control epilepsy.

  * uncontrolled epilepsy is defined as: more than 1 generalized seizure in any month within the 3 months prior to the day 1 visit, or
  * history of any of the following within 9 months prior to the day 1 visit: prolonged seizures or repetitive seizure activity requiring administration of a rescue benzodiazepine (oral, rectal, etc.) more than once a month, seizures lasting more than 10 minutes, status epilepticus or epilepsy with autonomic involvement.
* Concurrent participation in other therapies or interventions for autism during the
* study period and within the last 6 months.
* Logistical or situational limitations that prevent regular attendance at treatment
* sessions.
* History of significant adverse reactions to similar treatments or involving the use of anesthesia.
* Presence of serious behavioral problems or aggression that may affect the safety of the subject or staff during treatment sessions.
* Current or recent (previous 14 days) history of clinically significant bacterial, fungal, viral or mycobacterial infection.
* Presence of implanted medical devices or metallic foreign bodies that are not compatible with magnetic resonance imaging (MRI) or with the NeuroCytotron device, including but not limited to pacemakers, cochlear implants, deep brain stimulators, spinal cord stimulators, or any ferromagnetic implants.
* Participants diagnosed with ASD will be excluded from the protocol if they present any of the following conditions identified through imaging studies:
* Major Structural Lesions:
* Primary or metastatic brain tumors that compromise general neurological function.
* High-Risk Vascular Abnormalities:
* Arteriovenous malformations or aneurysms with an immediate risk of rupture or bleeding.
* Evidence of Acute Neurological Damage:
* Recent cerebral infarction (< 3 months).
* Active intracranial hemorrhage.
* Pathologies Interfering with Outcome Assessment:
* Severe cerebral atrophy that significantly impacts the likelihood of response to treatment.
* Severe congenital brain anomalies unrelated to the primary diagnosis of autism.
* Active Pathologies Incompatible with the Protocol:
* Intracranial infections, abscesses, or any evidence of active inflammation seen in imaging studies.

Ages: 3 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 256 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2029-02-01 (Estimated); Study Completion 2029-05-29 (Estimated)

PRIMARY OUTCOMES:
Change in Autism Diagnostic Observation Schedule, Second Edition (ADOS-2) total score | Baseline (pre-treatment, Days -3 to -1) to 12 weeks after the end of treatment
  ADOS-2 is a standardized, semi-structured assessment that measures social communication, interaction, play, and restricted or repetitive behaviors in individuals with autism spectrum disorder. Higher total scores indicate greater severity of ASD symptoms. The primary outcome is the change in ADOS-2 total score from baseline to 12 weeks post-treatment, comparing participants treated with NeuroCytotron functional neurogenesis stimulation therapy to those treated with placebo. A decrease in score reflects improvement in core ASD symptoms.

SECONDARY OUTCOMES:
Change in Childhood Autism Rating Scale, Third Edition (CARS-3) total score | Baseline (pre-treatment, Days -3 to -1) to 12 weeks after the end of treatment
  The CARS-3 is a clinician-rated scale with 15 items that assess autism symptom severity based on direct observation. Each item is rated from 1 (within normal limits) to 4 (severely abnormal); total scores range from 15 to 60, with higher scores indicating more severe symptoms of autism. The secondary outcome will be the change in CARS-3 total score from baseline to 12 weeks post-treatment, comparing the NeuroCytotron and placebo groups. A decrease in score reflects improvement in autism severity.
Incidence and severity of treatment-emergent adverse events and serious adverse events | From first treatment session (Day 1) through 12-week follow-up (approximately 14 weeks total per participant)
  Adverse events (AEs) are any untoward medical occurrences in a participant, whether or not related to the investigational device. Serious adverse events (SAEs) include events that result in death, are life-threatening, require or prolong hospitalization, cause significant disability, or are otherwise medically significant. The outcome will summarize the number and percentage of participants with AEs, SAEs, and AEs leading to discontinuation in each group, as well as severity and relationship to study treatment, and overall tolerability based on caregiver/participant reports collected at each visit.
Change in Gilliam Autism Rating Scale, Third Edition (GARS-3) total score | Baseline to 12 weeks after the end of treatment
  GARS-3 is a standardized rating scale used to identify and assess autism in individuals aged 3 to 22 years. It includes subscales for Social Interaction, Communication, and Stereotyped Behaviors, which contribute to a total score; higher scores indicate a greater likelihood or severity of autism. The secondary outcome is the change in GARS-3 total score from baseline to 12 weeks post-treatment, with lower scores indicating reduced autism-related behaviors, compared between treatment groups.
Change in Adaptive Behavior Assessment System, Third Edition (ABAS-3) composite score | Baseline to 12 weeks after the end of treatment
  ABAS-3 is a caregiver- or teacher-completed questionnaire that evaluates adaptive functioning across multiple domains (communication, community use, functional academics, home living, health and safety, leisure, self-care, self-direction, social, and work). Higher scores indicate better adaptive functioning. The secondary outcome will be the change in ABAS-3 composite score from baseline to 12 weeks post-treatment, with higher post-treatment scores reflecting improvement, compared between treatment groups.

OTHER OUTCOMES:
Change in brain regional volumes on structural MRI | Baseline (pre-treatment) to 12 weeks after the end of treatment
  High-resolution structural MRI will be used to quantify the volumes of gray and white matter in cortical, subcortical, and cerebellar regions (e.g., total cortical gray matter, cerebral white matter, thalamus, basal ganglia, hippocampus, amygdala, brainstem, and cerebellum). The exploratory outcome will compare within-subject and between-group changes in regional brain volumes from baseline to 12 weeks post-treatment for NeuroCytotron versus placebo. Increases in gray matter or cerebellar volumes and/or reductions in ventricular volume will be explored as potential markers of structural plasticity associated with treatment.
Change in white matter integrity on diffusion tensor imaging (DTI) | Baseline to 12 weeks after the end of treatment
  Diffusion tensor imaging will be used to assess white matter integrity using metrics such as fractional anisotropy (FA) and mean diffusivity (MD) in major white matter tracts related to cognitive and sensorimotor functions. Tract-based and connectome analyses will examine changes in FA, MD, and streamline counts between baseline and 12 weeks post-treatment. This exploratory outcome will compare changes in these DTI metrics between NeuroCytotron and placebo groups as potential indicators of treatment-related changes in structural connectivity.
Change in EEG spectral power, connectivity, and event-related potentials | Baseline, end of treatment (Day 28), and 4, 8, and 12 weeks after the end of treatment
  Resting-state EEG will be recorded using a 19-channel 10-20 system at baseline, after the last treatment session (Day 28), and during follow-up visits. Exploratory analyses will include (1) spectral power in standard frequency bands (delta, theta, alpha, beta); (2) functional connectivity metrics such as coherence and phase synchronization between key regions (e.g., frontal-parietal, fronto-temporal); and (3) event-related potentials (e.g., P300, N200) where applicable. The outcome will describe within-subject trajectories and between-group differences in these EEG measures over time as potential biomarkers of neurophysiological response to NeuroCytotron versus placebo.
Change in comorbid symptoms (anxiety, depression, sleep) and sensory processing difficulties | Baseline to 12 weeks after the end of treatment
  Exploratory outcomes will include changes in comorbid symptoms commonly associated with ASD-such as anxiety, depressive symptoms, and sleep disturbances-plus changes in sensory processing difficulties (hypersensitivity or hyposensitivity). These domains will be assessed with caregiver-reported standardized questionnaires, including sensory processing tools such as the Sensory Profile. Changes in questionnaire scores from baseline to 12 weeks post-treatment will be summarized and compared between the NeuroCytotron and placebo groups to explore broader functional effects of treatment beyond core ASD symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Jose R Trujillo, M.D., Sc.D., Study Chair — Neurocytonix, Inc.; Lorenzo R Morales Mancias, M.D., Principal Investigator — Neurocytonix, Inc.
Locations (2):
- NeuroCytonix, Inc., Rockville, Maryland, United States
- NeuroCytonix Mexico, San Pedro Garza García, Nuevo León, Mexico

IPD SHARING:
Plan to Share IPD: Undecided